CLINICAL TRIAL: NCT01247259
Title: Efficacy of Sublingual Immunotherapy With House Dust Mite Extract in Poly-allergen-sensitized Allergic Rhinitis Patients
Brief Title: Efficacy of Sublingual Immunotherapy in Polysensitized Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLIT-POLYSENSITIZATION
Record Dates: First submitted 2010-11-18; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; immunotherapy; sublingual
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLIT-mono (Active Comparator)
  Interventions: Drug: Pangramin®
- SLIT-poly (Active Comparator)
  Interventions: Drug: Pangramin®

INTERVENTIONS:
Drug: Pangramin® — During a 4-week increasing-dose phase, the patients increased the daily dose from 1 to 5 drops of 1.6 STU/mL solution from day 1 to 10, 1 to 5 drops of 8 STU/mL solution from day 11 to 15, 1 to 5 drops of 40 STU/mL solution from day 16 to 20, 1 to 5 drops of 200 STU/mL solution from day 21 to 25, and 1 to 5 drops of 1000 STU/mL solution from day 26 to 30. After reaching the maintenance dose, 5 drops of 1000 STU/mL solution, the patients took the allergen three times per week during the maintenance phase.

SUMMARY:
Recently, interest has increased in sublingual immunotherapy (SLIT) for treating allergic rhinitis. It is often suggested that polysensitized patients might not benefit from specific immunotherapy as much as monosensitized patients, although further research on this subject is needed. This study compared the efficacy of SLIT with standardized house dust mite extract in mono- and polysensitized allergic rhinitis patients.

Patients who were sensitized to house dust mites and treated with SLIT for house dust mites for at least 1 year between November 2007 and March 2010 were included. The mono-allergen sensitized group (Mgr) was defined as the patients who were sensitized to Dermatophagoides pteronyssinus (Dp) or D. farinae (Df; n = 70). The poly-allergen sensitized group (Pgr) was defined as the patients who were simultaneously sensitized to house dust mites and other allergens (n = 64). A standardized extract of house dust mites was used for immunotherapy. Anti-allergic medication and the total nasal symptom score (TNSS), including rhinorrhea, sneezing, nasal obstruction, and itchy nose, were evaluated before and 1 year after SLIT.

This study enrolled 134 patients. The TNSS improved significantly after SLIT in both groups, while the change in the TNSS did not differ significantly between the groups. The anti-allergic medication scores also decreased significantly in both groups, but there was no significant difference between the groups.

In polysensitized allergic rhinitis patients, SLIT for Dp/Df gave comparable improvements in both nasal symptoms and rescue medication scores to those in monosensitized patients, regardless of other positive allergens. SLIT for Dp/Df might be considered in polysensitized allergic rhinitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had sneezing, itching, rhinorrhea, and nasal congestion with or without eye symptoms
* patients who were sensitized to Dermatophagoides pteronyssinus (Dp) or D. farinae (Df), as confirmed by skin prick testing (A/H ratio ≥ 1) or MAST

Exclusion Criteria:

* Patients who had immunotherapy in the preceding 3 years
* Patients who had systemic immunological disorders

Ages: 4 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
total nasal symptom score (TNSS) and anti-allergic medication score (AMS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Young Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Otorhinolaryngology, Seoul National University Hospital, Seoul, South Korea